CLINICAL TRIAL: NCT06205875
Title: High Versus Low Dose Serratus Anterior Plane Block After Minimally Invasive Valve Surgery: a Double-blinded Randomized Controlled Trial.
Brief Title: High Versus Low Dose Serratus Anterior Plane Block After Minimally Invasive Valve Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principle investigator, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: f/2023/119
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Analgesia; Surgery; Cardiac Disease; Post Operative Pain
Keywords: Aorta/mitral valve surgery; Serratus anterior plane block; Enhanced recovery after surgery; post operative pain
MeSH Terms: conditions — Agnosia; Heart Diseases; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: This trial is designed as a mono-center, double-blinded, prospective, randomized controlled superiority trail comparing 2 groups of patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will receive a mixture of high-dose local anesthetic and epinephrine administered via a serratus anterior plane block.
  Interventions: Procedure: High dose serratus anterior plane block (2.4 mg/kg patient ideal body weight); Drug: PCIA with morphine
- Control group (Active Comparator): Patients in the control group will receive a serratus anterior plane block with a low dose local anesthetic (based upon our primary trial).
  Interventions: Procedure: Low dose serratus anterior plane block (1.2mg/kg patient ideal body weight); Drug: PCIA with morphine

INTERVENTIONS:
Procedure: High dose serratus anterior plane block (2.4 mg/kg patient ideal body weight) — The needle will be introduced in-plane from supero-anterior to postero-inferior until the needle tip is positioned in the plane underneath the serratus muscle (deep compartment). Under continuous ultrasound guidance, 3/4th of the bupivacaine 0.25% plus epinephrine solution will be injected in the deep compartment. After the deep component of the serratus anterior plane block is completed, the needle will be withdrawn to the subcutaneous tissues. The needle will be flattened and advanced in-plane to the plane superficial to the serratus muscles. The remainder quarter of the bupivacaine 0.25% plus epinephrine solution will be injected superficial to the serratus muscles after correct placement of the needle tip is confirmed on ultrasound. In total a dose of 2.4mg/kg patient ideal body weight will be administered. There is a maximal dose of 200 mg adrenalized bupivacaine for patients with an ideal body weight of 83 kg or more.
  Arms: Intervention group
Procedure: Low dose serratus anterior plane block (1.2mg/kg patient ideal body weight) — The needle will be introduced in-plane from supero-anterior to postero-inferior until the needle tip is positioned in the plane underneath the serratus muscle (deep compartment). Under continuous ultrasound guidance, 3/4th of the bupivacaine 0.25% will be injected in the deep compartment. After the deep component of the serratus anterior plane block is completed, the needle will be withdrawn to the subcutaneous tissues. The needle will be flattened and advanced in-plane to the plane superficial to the serratus muscles. The remainder quarter of the bupivacaine 0.25% will be injected superficial to the serratus muscles after correct placement of the needle tip is confirmed on ultrasound.
  Arms: Control group
Drug: PCIA with morphine — A patient controlled intravenous analgesia system (Bodyguard 595 Colorvision®) with morphine (Sterop®) using following settings: bolus 1.5 mg and lockout interval 7 min with maximal dose of 30mg per 4 hours.
  Other Names: PCIA with Sterop

SUMMARY:
This study aims to compare the efficacy and quality of pain relief provided by the high-dose serratus anterior plane (SAP) block with the standard SAP block in preventing and treating acute postoperative pain after total endoscopic aortic or mitral valve surgery.

DETAILED DESCRIPTION:
During the last two decades, cardiac surgical techniques have changed dramatically. Evidence for good short and long-term outcomes after endovascular and minimally invasive procedures is rising. This shift made it possible to avoid sternotomy and thus facilitating earlier patient recovery without compromising safety. Therefore, enhanced recovery after surgery (ERAS) protocols have been implemented to aim for early extubation and ambulation. While policies for early extubation and discharge from the hospital have been implemented, the analgesic regimen has not been modified. Opioids remain the standard treatment in the postoperative setting after cardiac surgery despite known side effects such as nausea, constipation and the risk of addiction. Neuraxial anaesthesia techniques, which require fewer opioids in cardiac surgery, have been studied and validated but not yet implemented.

In 2013, the serratus anterior plane (SAP) block was described as a pain relief option for chest surgery. This anaesthesia technique injects local anaesthetics under the serratus muscle and between the latissimus dorsi and serratus anterior using ultrasound. Successful pain relief with this SAP block has been reported in thoracotomy, chest surgery, and rib fractures. In our previous study, we demonstrated a 40% reduction in morphine consumption during the first 24 hours after total endoscopic aortic valve replacement with an SAP block compared to a control group without an SAP block. Lower pain scores were also observed in the SAP group

As such, in this proposed study, we aim to optimise the intensity of the Serratus anterior plane block (SAPB) to decrease opioid requirements further and to encounter more favourable secondary clinical outcome parameters. One strategy to increase the duration of action of plane blocks is injecting higher doses of local anaesthetics. A meta-analysis by De Oliveira et al. on transabdominal plane (TAP)-blocks for abdominal surgery showed a correlation between the local anaesthetic dose and the late block effect, impacting both pain scores and opioid consumption. In a randomised controlled trial by Suresh, a TAP block with bupivacaine 1.25 mcg/kg was compared to a TAP block with bupivacaine 2.5 mcg/kg, revealing a longer duration of analgesia and a lower need for additional analgesics up to 24 hours post-surgery. Moreover, loading doses up to 2mg/kg body weight are recommended for truncal blocks in general, but the mean injected dose in our intervention group was 1.25mg/kg, considering a mean patient body weight of 79.2kg. Notably, a pharmacokinetic study by Maximos and colleagues on an adrenalised bupivacaine mixture after pectointercostal fascial plane block (PIFB) after cardiac surgery showed that, despite injecting 2mcg/kg adrenalised bupivacain, both total and free arterial serum bupivacaine levels were 10-20 times lower than levels associated with neurologic or cardiovascular toxicity in the literature.

In conclusion, we are convinced we can safely improve the late effects of our SAPB compared to our first study by increasing the dose of the local anesthetic injectate.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective aortic valve surgery or elective mitral valve surgery via right anterolateral thoracotomy
* Adult patients (minimally 18 years old)
* Bodyweight > 50kg
* EuroScore ii < 3%

Exclusion Criteria:

* Refusal to participate
* Inability to communicate due to language or neurologic barriers
* Inability to control and self-administer opioids with PCIA or to comprehend the NRS pain score due to confusion or learning difficulties
* Chronic use of opioids
* Chronic use of analgesic antidepressants and/or antiepileptics
* Use of prohibited medication which possibly interacts with bupivacaine-epinephrine or opioids (mexiletine, ketoconazole, theophylline, IMAO, Digitalis and cimetidine)
* History of major trauma or surgery to right chest wall
* History of chronic pain at right chest wall
* Allergy to opioids and/or local anesthetics
* Allergy to paracetamol
* Class 3 obesity (BMI 40 or more)
* Pregnancy
* Intraoperative events compromising early postoperative recovery (aortic dissection, systolic anterior motion of the mitral valve, cardiac tamponade, brady-arrhytmias requiring external pacing,...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption by patient-controlled intravenous analgesia (PCIA) | 24 hours after block placement
  Morphine consumption will be directly read from the PCIA-system after 24 hours

SECONDARY OUTCOMES:
Opioid consumption during predetermined time intervals after surgery | Every 4 hours until 24 hours after placement of the SAP block
  Morphine consumption will be directly read from PCIA-system at predetermined time intervals after performing the SAP block.
Opioid free patients first 24 postoperative hours | First 24 hours
  Number of patients that do not require any additional opioids within the first 24 hours after block placement.
Postoperative pain score in rest and on deep respiration | 4, 8, 12 and 24 hours after performing the SAP block and at postoperative day 7.
  The postoperative pain in rest, as well as with deep respiration on the surgical site, is evaluated based on an 11-point numeric scale (NRS) where 0 = no pain and 10 = worst pain ever.
Overall patient Satisfaction with analgesic therapy | 24 hours after performing the SAP block at postoperative day 1.
  Overall patient satisfaction with analgesic therapy will be assessed with an 11-point NRS scale (where 0 = not satisfied at all and 10 = extremely satisfied)
Time to extubation | Throughout study completion, an average of 7 days
  Time from arrival to the ICU until extubation in minutes.
Time to first mobilization | Intended at 6 hours after surgery
  Time from arrival to the ICU until first mobilization.
Postoperative nausea and vomiting (PONV) | 24 hours after performing the SAP block at postoperative day 1
  The simplified PONV impact scale will be used to asses PONV. Clinically important PONV will be defined as a score of 5 or more.
Constipation | Until postoperative day 7
  Time to first defecation (postoperative days) or need for laxatives during hospital stay (number of patients)
ICU length of stay | Until postoperative day 7
  Time from arrival to the ICU until meeting discharge criteria to the ward in postoperative hours.
Hospital length of stay | Throughout study completion, an average of 7 days
  Time to discharge out of the hospital in postoperative days (day of surgery = day 0)
Pneumonia | Until postoperative day 7
  Defined as empirical antibiotic therapy for suspicion of pneumonia during hospital stay, in number of patients.
Quality of recovery | At postoperative day 2 and 7
  Quality of recovery will be assessed with Quality of Life questionnaires: EuroQol*5D (EQ5D) and short form health survey (SF-36).
Bupivacaine dosage | at 30minutes as well as at 1, 2, 4 and 8 hours after block placement
  In the first 36 study patients, arterial blood samples will be taken to calculate the dosage of total and free plasma bupivacaine levels. For each patient 5 samples will be collected, with a total amount of 50 ml blood per patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No